CLINICAL TRIAL: NCT06920121
Title: Effects of Virtual Reality Glasses and Stress Ball on Distress and Pain During Arteriovenous Fistula Cannulation
Brief Title: Virtual Reality Glasses and Stress Ball on Distress and Pain Arteriovenous Fistula Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, Principal Investigator, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/08
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-07

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality glasses (Experimental): Virtual reality glasses Beginning 2-3 minute before the start of the procedure, the patients will be watched (5 minutes) with an android mobile phone inserted into the Cardboard Super Flex Binoculars Glasses, with a music background, licensed product.
  Interventions: Other: Virtual reality glasses
- Stress ball (Experimental): Before AVF cannulation, patients will be given a round, colored, medium-hard, high-quality silicone squeezable ball (the arm without vascular access will be used). In order to avoid implying that the procedure is inherently stressful, patients will be given the name squeeze ball when they are given information about the stress ball application. Patients will be instructed to continue squeezing and relaxing the stress ball (squeezing and relaxing once, counting from one to three) for 5 minutes before and throughout the AVF cannulation procedure. Patients will be instructed to focus their attention on the stress ball and focus on squeezing the stress ball.
  Interventions: Other: Stress ball
- Control grups (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Virtual reality glasses — Virtual reality glasses Beginning 2-3 minute before the start of the procedure, the patients will be watched (5 minutes) with an android mobile phone inserted into the Cardboard Super Flex Binoculars Glasses, with a music background, licensed product.
  Arms: Virtual reality glasses
Other: Stress ball — Patients will be instructed to continue squeezing and relaxing the stress ball (squeezing and relaxing once, counting from one to three) for 5 minutes before and throughout the AVF cannulation procedure. Patients will be instructed to focus their attention on the stress ball and focus on squeezing the stress ball.
  Arms: Stress ball

SUMMARY:
Effects of Virtual Reality Glasses and Stress Ball on Distress and Pain During Arteriovenous Fistula Cannulation. The research was conducted as a randomized experimental study with a pre-test - post-test control group.

DETAILED DESCRIPTION:
Beginning 1-2 minute before the start of the procedure, the patients will be watched (5 minutes) with an android mobile phone inserted into the Cardboard Super Flex Binoculars Glasses.

A stress ball will be applied to the patient 1-2 minutes before the start of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old,
* Be able to speak and understand Turkish,
* Have the cognitive ability to answer the data collection tools,
* Be willing to participate in the study,
* Participate in a hemodialysis program three days a week,

Exclusion Criteria:

* Having a communication problem (hearing, language, understanding, etc.),
* Having a psychiatric diagnosis (To be checked from medical records),
* Having failed AVF cannulation at the first attempt,
* Having any signs of infection such as redness, swelling, open wound in the area where the procedure will be performed,
* Having used a sedative within the last 8 hours,
* Having used any painkillers before the procedure on the same day,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline, pre-intervention (Before AVF cannulation procedure)
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. VAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
Visual Analog Scale | Immediately after the intervention (After AVF cannulation procedure)
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. VAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
The Distress Thermometer (DT | Baseline, pre-intervention (Before AVF cannulation procedure)
  The Distress Thermometer is a scale developed by Roth et al. (1998) for determining psychological distress in cancer patients. The thermometer is a Likert-type scale with scores from 0 (no stress) to 10 (excessive stress). In a short and easy-tounderstand scale, patients can easily mark their distress levels in ranges indicated on the thermometer. The Turkish validity-reliability study of the Distress Thermometer for cancer patients was performed by Özalp et al. and the recommended cut-off score for the thermometer in this study was set at four and above.
The Distress Thermometer (DT | Immediately after the intervention (After AVF cannulation procedure)
  The Distress Thermometer is a scale developed by Roth et al. (1998) for determining psychological distress in cancer patients. The thermometer is a Likert-type scale with scores from 0 (no stress) to 10 (excessive stress). In a short and easy-tounderstand scale, patients can easily mark their distress levels in ranges indicated on the thermometer. The Turkish validity-reliability study of the Distress Thermometer for cancer patients was performed by Özalp et al. and the recommended cut-off score for the thermometer in this study was set at four and above.

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz Özer, Principal Investigator — İstanbul Sabahattin Zaim Üniversitesi
Locations (1):
- Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Küçükçekmece, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toraman RL, Eskici Ilgin V. Effect of Virtual Reality Glasses Application on Pain, Anxiety, and Patient Satisfaction During a Transrectal Prostate Biopsy: A Randomized Controlled Trial. Biol Res Nurs. 2024 Oct;26(4):485-497. doi: 10.1177/10998004241236154. Epub 2024 Feb 28. PMID 38418943